CLINICAL TRIAL: NCT02109952
Title: The Purpose of This Study is to Monitor Fracture Risk Associated With Bone Tumors in Cancer Patients
Brief Title: Biomechanics of Metastatic Defects in Bone
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ara Nazarian, Assistant Professor of Orthopedic Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000285
Record Dates: First submitted 2014-03-31; First posted 2014-04-10 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer Bone; Bone Tumors
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to monitor fracture risk associated with bone tumors in cancer patients.

Previous studies from our lab have suggested that it is possible to compute the mechanical strength of bones with tumors using computed tomography (CT) scans, which are like three-dimensional X-ray pictures of the affected bones.

The next step in determining the usefulness of this type of strength analysis is to see if we can accurately predict who is at risk for bone fracture and which patients are at high risk of fractures.

This non-invasive analysis may help physicians determine the best treatment to reduce the risk of an impending bone fracture in the future.

DETAILED DESCRIPTION:
If a patient agrees to participate in this study, we will ask the patient to complete two written, self-administered questionnaires. The questionnaires will take about fifteen minutes to complete and contain questions about the patient's general health as well as questions specific to the site of the bone tumor. The patient will be asked to complete the first questionnaire upon enrollment in the study, and the second when participation in the study is concluded. The patient will be asked to complete and return the questionnaire to the project coordinator at this time. If for any reason the patient is unable to complete the questionnaire at this time, he/she will be asked to return it to the project coordinator within two weeks using a stamped, pre-addressed envelope, which will be provided.

The treating physician has ordered both an X-ray picture and a three-dimensional CT scan image of the involved bone plus the contralateral limb (lower limbs). He/she will be provided with a standard report from the radiologist describing the appearance of the bone tumor and the bone itself which the treating physician will use to determine the course of treatment he/she deems appropriate. We will perform a special analysis of the CT images that will allow us to estimate the strength of the bone with the tumor. Based on this engineering analysis of the strength of the bone, the treating physician may alter the prescribed treatment to decrease the risk that bone will fracture. If the patient does not have a fracture within the follow-up period (four months), he/she will undergo a second CT scan to determine the response of the tumor to treatment and changes in the strength of the bone. If the patient does have a fracture within the follow-up period, he/she will undergo a second CT scan to determine the integrity of the remaining bone to help your physician plan the next course of action. We will use the second CT scan to estimate how weak the bone was just prior to fracture. In either case, the patient's participation in this study will be concluded after the second CT scan.

Patient participation in the study will last four months. If the patient has a fracture before four months, his/her participation will end at that time.

The investigator and/or the treating physician may decide to take the patient off this study if

1. patient refuses or is unable to complete study procedures;
2. patient develops weakness or numbness in his/her limbs due to your disease;
3. patient's bone fractures due to significant trauma (e.g., traffic accident, fall from height);
4. a different bone fractures, limiting patient's ability to put pressure on the bone of interest; or
5. patient relocate.

The patient can end his/her participation at any time. The patient's decision to withdraw from the study will not affect in any way his/her medical care and/or benefits. If the patient decides to end his/her participation in the study, we encourage him/her to discuss the decision the treating physician.

STUDY LOCATION Privacy Patients will be approached by treating physicians at clinic and privately (in the examination room), where they can privately describe the study, answer any questions the patient might have and potentially enroll the patient in the study. Patient privacy and confidentiality will be strictly observed during all steps of recruitment, reporting of data and follow up conversations.

Physical Setting

All patient related activity will be conducted in the hospital as the patient undergoes treatment. CT data analysis will be performed at the Center for advanced Orthopaedic Studies at BIDMC.

DATA SECURITY All data will be kept behind BIDMC firewall at an access controlled computer designated for this study only. Additionally, the patient data will be anonymized and a number will be assigned to protect the patient identity, therefore those conducting analysis on the CT data will have no access to patient identifiable information.

ELIGIBILITY:
Inclusion Criteria:

Patient with metastatic cancer bone lesions

Exclusion Criteria:

-

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: When a patient presents to the orthopaedic oncologist with lower appendicular skeletal skeletal metastasis, as per standard clinical practice biplanar radiographs and CT scans of the involved bone(s) plus the contralateral limb will be obtained. Informed consent will be obtained for CT scan with the contralateral limb (Both limbs are in the gantry and are imaged together-this is not an additional step, as this is how patients are scanned for general care of lesions in the lower limbs) to provide a patient specific internal control and calcium hydroxyapatite phantom for standardizing bone density estimates. Post-processing of the image data will be conducted by the Orthopaedic Biomechanics Lab at BIDMC to calculate fracture risk associated with the bone lesion.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2009-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fracture Risk Assessment in Patients with Skeletal Metastasis | 0-4 Months
  Based on past studies, metastatic lesion in cancer bone alters both the material and geometric properties of the bone while rigidity, the structural property, integrates both two properties in bone. For a cancerous bone, the axial (EA), bending (EI), and torsional (GJ) rigidity determine the capacity of the bone to resist axial, bending and twisting loads respectively. Because the weakest segment of the bone dictates the load capacity of the entire bone, we have developed algorithms to calculate the minimal rigidity of a bone with an osteolytic lesion using serial, trans-axial, computed tomography (CT) images through the affected bone to measure both the bone tissue mineral density and cross-sectional geometry. If the ratio of EA, EI or GI in compare with the normal bone's EA, EI, or GI was 65% or less, pathological fracture will be predicted. This non-invasive analysis may help physicians determine the best treatment to reduce the risk of an impending bone fracture in the future.

SECONDARY OUTCOMES:
Fracture Risk Assessment in Patients with Skeletal Metastasis (Following-up with Changes) | 4-12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ara Nazarian, PhD, Principal Investigator — anazaria@bidmc.harvard.edu
Locations (8):
- United States (7):
  - Alvin and Lois Lapidus Cancer Center, Sinai Hospital of Baltimore, Inc, Baltimore, Maryland
  - Department of Orthopaedic Surgery, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - Department of Orthopaedic Surgery, University of Minnesota Medical Center, Minneapolis, Minnesota
  - Department of Orthopedic Surgery, Upstate Medical University, Syracuse, New York
  - Department of Orthopaedic Surgery, Rhode Island Hospital, Providence, Rhode Island
  - Section of Orthopaedic Oncology, University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Edwards Comprehensive Cancer Center, Marshall University, Huntington, West Virginia
- Department of Orthopaedic Surgery, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- See also: Guide website to join this study — http://www.bidmc.org/Research/Departments/Orthopaedic-Surgery/NazarianLab/MSTS.aspx